CLINICAL TRIAL: NCT05696223
Title: Doppler at the Diagnosis in Predicting Perinatal Outcomes in Early and Late-onset Fetal Growth Restriction
Status: Completed | Type: Observational
Sponsor: Central Hospital, Nancy, France (Other)
Responsible Party: Principal Investigator, TOURNIER Mathilde, Doctor, Central Hospital, Nancy, France
Other Study IDs: 2022PI187-343
Record Dates: First submitted 2023-01-13; First posted 2023-01-25 (Actual); Last update posted 2023-01-25 (Actual); Status verified 2023-01

CONDITIONS: Fetal Growth Retardation
Keywords: Fetal Growth Retardation, Doppler, perinatale outcome
MeSH Terms: conditions — Fetal Growth Retardation | interventions — High-Energy Shock Waves

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Early fetal growth restriction: Fetal growth restriction diagnosed before 32 SA
  Interventions: Other: Ultrasound
- Late fetal growth restriction: Fetal growth restriction diagnosed after 32 SA
  Interventions: Other: Ultrasound

INTERVENTIONS:
Other: Ultrasound — Doppler mesure

SUMMARY:
When a FGR is diagnose, the challenge in his monitoring is to assess the benefit-risk balance between continuing the pregnancy in order to limit complications related to prematurity and birth in order to minimize any risk of fetal death in utero. By able to know the characteristics of fetal deteriorations and its relationship with fetal and neonatal outcomes could be a thankful help in this decision. The placental insufficiency is by far the most common cause of FGR (32)(miller 2008). This effect can be documented thanks to ultrasound examinations to study fetal growth and Doppler of umbilical arteries for the placenta, the middle cerebral artery for the brain perfusion and the Ductus Venosus for the cardiac effects of placental dysfunction. The apparition of Doppler abnormalities suggests a deterioration of the disease and leads to several changes in clinical FGR management. Nevertheless, at this time, very few studies allow us to predict the time util the degradation and their impact on perinatal outcomes.

The primary aim of this study was to evaluate the performance of the Doppler at the time of diagnosis in predicting the outcome of pregnancies. The secondary aim was to evaluate the performance of Doppler performed at any time during pregnancy and studied independently in predicting outcome of pregnancies

ELIGIBILITY:
Inclusion Criteria:

* Fetal growth restriction of antenatal diagnosis

Exclusion Criteria:

* Twin pregnancies, non-isolated IUGR, post-natal diagnosis of FGR and incomplete records

Ages: 18 Years to 50 Years | Sex: Female
Age Groups: Adult
Study Population: All the FGR of antenatal diagnosis, who were confirmed by an ultrasound made by a referring Doctor and involved in a specific management for FGR, during this period of 2 years were included
Sampling Method: Non-Probability Sample
Enrollment: 220 (Actual)
Dates: Start 2022-06-01 (Actual); Primary Completion 2022-12-01 (Actual); Study Completion 2023-01-01 (Actual)

PRIMARY OUTCOMES:
evaluate the performance of the Doppler at the time of diagnosis in predicting the outcome of pregnancies | during pregnancy (6 month per patient maximum)

SECONDARY OUTCOMES:
evaluate the performance of Doppler performed at any time during pregnancy and studied independently in predicting outcome of pregnancies | during pregnancy (6 month per patient maximum)

CONTACTS AND LOCATIONS:
Locations (1):
- Maternite Regionale et Universitaire de Nancy, Nancy, Meurthe-et-moselle, France

IPD SHARING:
Plan to Share IPD: No